CLINICAL TRIAL: NCT06731179
Title: STUDY TO EVALUATE THE ROLE OF T CELL-DYSFUNCTION IN SYMPTOMS ASSOCIATED WITH LONG COVID, LYME DISEASE AND MYALGIC ENCEPHALOMYELITIS/CHRONIC FATIGUE SYNDROME USING THE VIRAXIMMUNE FLUOROSPOT T CELL ASSAY
Brief Title: A Prospective Study to Evaluate the Role of T-Cell Dysfunction in Patients Who Present Symptoms Associated With Long COVID, Lyme Disease and Myalic Encephalomyelitis / Chronic Fatigue Syndrome Using the Vira Immune Fluorospot T Cell Assay
Status: Active, not recruiting | Type: Observational
Sponsor: ViraxBio Labs (Network)
Responsible Party: Sponsor
Other Study IDs: VRX - 002
Record Dates: First submitted 2024-12-11; First posted 2024-12-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-03

CONDITIONS: Long COVID; PTLDs; Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) (ICD-10 G93.3)
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Residual blood specimens - frozen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Long COVID diagnosis: Long COVID diagnosis
- ME/CFS symptoms: ME/CFS symptoms
- PTLDS symptoms: PTLDS symptoms
- Healthy Individuals: Healthy Individuals

SUMMARY:
This is a longitudinal observational study recruiting individuals that have attended three clinical sites with symptoms associated with a diagnosis of long COVID, PTLDS or ME/CFS. The study will be a multi-centre study, with up to 160 male and female participants enrolled. Participants that experience symptoms considered to be associated with a diagnosis of long COVID, PTLDS or ME/CFS will consent to the study, and attend for two study visits (at study entry and 6 months) to complete a questionnaire related to their symptoms, and to have a blood sample taken. Blood samples will be taken either at the clinical site or at the participant's home if they are unable to attend due to the severity of their illness. . Participants will be allocated to one of the following groups:

Group 1: Long COVID Group 2: ME/CFS Group 3: PTLDS Group 4: Healthy Control

ELIGIBILITY:
Persistent symptoms for groups 1-3 for consistency.

Inclusion Criteria:

1. Aged 18 years or older
2. History of acute COVID-19 infection (medically recorded)
3. Symptoms of fatigue and, shortness of breath and/or, joint pain and/or, problems with memory and concentration which have been present for more than a period of 6 months post infection
4. Nonsteroidal anti-inflammatory drugs (NSAIDs such as ibuprofen, diclofenac, aspirin, etc.) must have been stopped at least 48 hours prior to admission to the clinical research centre (evaluation through questionnaire).
5. Willing and able to sign the ICF and comply with study procedures.

Exclusion Criteria:

1. Taking immunosuppressive medication (including corticosteroids), or receiving chemotherapy, cytokine or anti-cytokine therapy, or antithrombotic medication (evaluation through questionnaire).
2. Significant and/or acute illness within 5 days prior to admission that may impact safety assessments, in the opinion of the Investigator.
3. Participants who are, in the opinion of the Investigator, not suitable for enrolment for another reason. For example, participants with: cognitive impairment or severe mental health conditions that might affect their ability to provide informed consent or follow study procedures; non-adherence risk where participants are unlikely to follow study protocols; participants with other chronic inflammatory conditions not under investigation e.g. inflammatory bowel disease, COPD that may have immune profiles that differ from the study's intended populationI

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Up to 120 male and female participants identified as having persistent symptoms associated with a diagnosis of long COVID, PTLDS or ME/CFS. Additionally, up to 40 healthy male and female who have not been clinically diagnosed as having symptoms associated with long COVID, PTLDS or ME/CFS will be enrolled as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Performance of the ViraxImmune FluoroSpot T cell assay (PPA / NPA - predicted outcome) | 18 months
  To evaluate the performance of the ViraxImmune FluoroSpot T cell assay to identify T cell dysfunction in participants diagnosed with long COVID, post treatment Lyme disease (PTLD) and Myalgic Encephalomyelitis/Chronic Fatigue (ME/CFS)

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Monklands University Hospital, NHS, Airdrie
  - Glasgow and Clyde NHS, Glasgow
  - Raigmore Hospital, Inverness, Inverness

IPD SHARING:
Plan to Share IPD: No